CLINICAL TRIAL: NCT01723982
Title: A Randomised, Placebo-controlled, Double-blind, Parallel Groups, Multinational, Multicentre Trial Assessing the Effect of Barusiban Administered Subcutaneously on the Day of Transfer on Implantation and Pregnancy Rates in IVF/ICSI Patients
Brief Title: Barusiban Subcutaneously for Reducing Implantation Failure Due to Uterine Contractions
Acronym: BASIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000048; 2012-001622-10 (EudraCT Number)
Record Dates: First submitted 2012-10-05; First posted 2012-11-08 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — barusiban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A. FE 200440 (Experimental): Barusiban (FE 200440) Solution for Injection for Subcutaneous use
  Interventions: Drug: Barusiban (FE 200440)
- B. Placebo (Placebo Comparator): Placebo Solution for Injection for Subcutaneous use
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Barusiban (FE 200440)
  Arms: A. FE 200440
Drug: Placebo Comparator
  Arms: B. Placebo

SUMMARY:
This trial investigates the effects of FE 200440 compared to placebo on implantation rate in women undergoing IVF/ICSI treatment

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-37 years
* Women who have undergone 2-4 previous fresh in vitro fertilization (IVF) or intracytoplasmatic sperm injection (ICSI) cycles that all resulted in a negative βhCG test, despite transfer of at least one embryo/blastocyst of good quality
* Women who have in the current controlled ovarian stimulation cycle for IVF/ICSI followed the long Gonadotrophin Releasing Hormone (GnRH) agonist or GnRH antagonist protocol, received hCG for triggering of final follicular maturation and have undergone oocyte retrieval for IVF/ICSI with the purpose of fresh transfer
* Retrieval of at least 6 oocytes in the current controlled ovarian stimulation cycle
* Subjects should have at least one embryo of good quality available for transfer on day 3, or at least one good quality blastocyst available for transfer on day 5

Exclusion Criteria:

* A total of 6 or more controlled ovarian stimulation cycles for IVF/ICSI
* Abnormal karyotype
* Uterine pathology or hydrosalpinx
* Diagnosed with acquired or congenital thrombophilia disease

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 256 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Ongoing implantation rate | 10-11 weeks after embryo transfer

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 10-11 weeks after transfer
Implantation rate | 5-6 weeks after transfer
Clinical pregnancy rate | 5-6 weeks after transfer
Positive Beta Human Chorionic Gonadotrophin (βhCG) rate | 13-15 days after transfer
Serum barusiban concentration at the expected tmax | 30 min after 2nd IMP administration
Frequency and intensity of adverse events | Within 60 days of oocyte retrieval +1 day until 10 -11 weeks after embryo transfer
Frequency and intensity of injection site reactions | Immediately and 30 min after each administration of IMP

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (14):
- Australia (3):
  - Westmead Fertility Centre, Westmead, New South Wales
  - Monash IVF, Clayton, Victoria
  - Melbourne IVF, Melbourne, Victoria
- Belgium (2):
  - UZ Brussel, Brussels
  - AZ Jan Palfijn Gent AV, Ghent
- Clinique OVO, Montreal, Quebec, Canada
- ICF CUBE, Prague, Czechia
- nOvum, Warsaw, Poland
- Spain (6):
  - IVI Alicante, Alicante
  - Dexeus, Barcelona
  - IVI Madrid, Madrid
  - IVI Sevilla, Seville
  - IVI Valencia, Valencia
  - IVI Zaragoza, Zaragoza